CLINICAL TRIAL: NCT04508179
Title: A Phase 1, Placebo-controlled, Within-Cohort Randomized, Double-blind, Single and Multiple Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of 7HP349 in Normal Healthy Male Subjects
Brief Title: A Phase 1 SAD and MAD Study of the Safety, Tolerability and PK of 7HP349 in Normal Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 7 Hills Pharma, LLC (Industry)
Collaborators: Frontage Clinical Services, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7HP-101a
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: This study consists of three parts, Part A, Part B and Part C, which will be undertaken sequentially. Part A is a SAD study to determine the safety, tolerability and PK of 7HP349 in healthy male subjects, and to define the OPD. Part B is a MAD study to determine the safety, tolerability and PK of 7HP349 following up to 5 once daily oral doses in healthy male subjects. Part C is a crossover study to evaluate the effect of the fed or fasting prandial state on the single dose PK of 7HP349.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 7HP349 Capsules (Experimental): Part A: 7HP349 Capsules (5 cohorts); Part B: 7HP349 Capsules (2 cohorts); Part C: 7HP349 Capsules (3-period cross-over)
  Interventions: Drug: 7HP349 Single Ascending Dose; Drug: 7HP349 Multiple Ascending Dose; Drug: 7HP349 Food Effect
- Placebo Capsules (Placebo Comparator): Part A: Placebo Capsules (5 cohorts); Part B: Placebo Capsules (2 cohorts)
  Interventions: Drug: Placebo Single Ascending Dose; Drug: Placebo Multiple Ascending Dose

INTERVENTIONS:
Drug: 7HP349 Single Ascending Dose — Part A: 7HP349 Capsules, Single Ascending Dose (SAD)
  Other Names: 7HP349 SAD
  Arms: 7HP349 Capsules
Drug: 7HP349 Multiple Ascending Dose — Part B: 7HP349 Capsules, Multiple Ascending Dose (MAD)
  Other Names: 7HP349 MAD
  Arms: 7HP349 Capsules
Drug: Placebo Single Ascending Dose — Part A: Placebo Capsules, Single Ascending Dose (SAD)
  Other Names: Placebo SAD
  Arms: Placebo Capsules
Drug: Placebo Multiple Ascending Dose — Part B: Placebo Capsules, Multiple Ascending Dose (MAD)
  Other Names: Placebo MAD
  Arms: Placebo Capsules
Drug: 7HP349 Food Effect — Part C: 7HP349 Capsules, Food Effect
  Other Names: 7HP349 FE
  Arms: 7HP349 Capsules

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of 7HP349, an allosteric integrin activator, in healthy male subjects

DETAILED DESCRIPTION:
This first-in-human (FIH) study consists of a placebo-controlled, sequential, dose escalation study to determine the safety, tolerability and pharmacokinetics (PK) of 7HP349 following single and multiple oral dose administration to healthy male subjects, with a separate, open-label food effect cohort at the optimal pharmacokinetic dose (OPD). The study will be carried out in 3 parts.

Part A: This is a placebo-controlled, within-cohort randomized, double-blind, sequential, single ascending dose (SAD) escalation study to determine the safety, tolerability and PK of 7HP349 following administration of single oral doses in healthy male subjects, and to define the OPD of 7HP349.

Part B: This is a placebo-controlled, within-cohort randomized, double-blind, sequential, multiple ascending dose (MAD) escalation study to determine the safety, tolerability and PK of 7HP349 following up to 5 once daily oral doses in healthy male subjects.

Part C: This is a randomized, open label, two-treatment, three-period, crossover study to evaluate the effect of the fed or fasting prandial state on the single dose PK of 7HP349.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the ages of 18 and 45 years, inclusive
* Normal clinical chemistry, hepatic function, hematology, thyroid function
* Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight not less than 60 kg
* Agree to refrain from consuming products containing grapefruit, pomelo, star fruit or Seville oranges for at least 7 days before the first dose of study drug until the final discharge evaluation
* Positive immune status as defined in serum as measles, mumps, varicella-zoster viruses (VZR); Antibody Index (AI) ≥ 1.1, and positive Rubella: AI ≥ 1.0

Exclusion Criteria:

* Clinically significant history of disorders, infections or drug hypersensitivity as determined by the Investigator
* History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody
* Current treatment or treatment within 30 days with another investigational medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 7HP349 in healthy male subjects as assessed by incidence of treatment-emergent adverse events according to CTCAE v5.0 criteria | 17 days
  Safety assessments will include evaluation of incidence of treatment-emergent adverse events (AEs) according to CTCAE v5.0 criteria, including vital signs, resting electrocardiogram (ECG) parameters, standard hematology, chemistry, urinalysis and other tests

SECONDARY OUTCOMES:
Pharmacokinetics of 7HP349 in healthy male subjects as assessed by maximum plasma concentration (Cmax) towards determination of the optimal pharmacokinetic dose (OPD) | 17 days
  Determination of maximum plasma concentration (Cmax)
Pharmacokinetics of 7HP349 in healthy male subjects as assessed by plasma exposure (AUClast and/or AUCinf) towards determination of the optimal pharmacokinetic dose (OPD) | 17 days
  Determination of plasma exposure (AUClast and/or AUCinf)
Pharmacokinetics of 7HP349 in healthy male subjects as assessed by exposure in urine towards determination of the optimal pharmacokinetic dose (OPD) | 17 days
  Determination of exposure in urine
Pharmacokinetics of 7HP349 in healthy male subjects as assessed by renal clearance (CLr) towards determination of the optimal pharmacokinetic dose (OPD) | 17 days
  Determination of renal clearance (CLr)
Effect of food on the pharmacokinetics of 7HP349 in healthy male subjects as assessed by measurement of maximum plasma concentration (Cmax) in fed individuals | 28 days
  Fed prandial state, determination of maximum plasma concentration (Cmax)
Effect of food on the pharmacokinetics of 7HP349 in healthy male subjects as assessed by measurement of maximum plasma exposure (AUClast and/or AUCinf) in fed individuals | 28 days
  Fed prandial state, determination of plasma exposure (AUClast and/or AUCinf)
Effect of food on the pharmacokinetics of 7HP349 in healthy male subjects as assessed by measurement of maximum plasma concentration (Cmax) in fasted individuals | 28 days
  Fasted prandial state, determination of maximum plasma concentration (Cmax)
Effect of food on the pharmacokinetics of 7HP349 in healthy male subjects as assessed by measurement of maximum plasma exposure (AUClast and/or AUCinf) in fasted individuals | 28 days
  Fasted prandial state, determination of plasma exposure (AUClast and/or AUCinf)
Effect of food on the pharmacokinetics of 7HP349 in healthy male subjects as assessed by measurement of the Geometric Mean Ratio (GMR) of the maximum plasma concentration (Cmax) in fed vs. fasted individuals | 28 days
  Determination of Geometric Mean Ratio (GMR) of fed:fasted Cmax
Effect of food on the pharmacokinetics of 7HP349 in healthy male subjects as assessed by measurement of the Geometric Mean Ratio (GMR) of the plasma exposure (AUClast and/or AUCinf) in fed vs. fasted individuals | 28 days
  Determination of Geometric Mean Ratio (GMR) of fed:fasted AUClast and/or AUCinf

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided